CLINICAL TRIAL: NCT01758094
Title: Plasma RBP Levels in Patients With Idiopathic Hypogonadotrophic Hypogonadism
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, MD, Gulhane School of Medicine
Other Study IDs: 24122012
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism
Keywords: hypogonadism; Retinol binding globulin 4; Testosterone treatment
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypogonadotropic hypogonadism patients: Treatment naive 25 patients with idiopathic hypogonadotrophic hypogonadism
  Interventions: Drug: Sustanon 250 mg ampule (Testosterone esters)

INTERVENTIONS:
Drug: Sustanon 250 mg ampule (Testosterone esters) — Drug used for treatment of hypogonadism
  Other Names: No name

SUMMARY:
The aim of the present study was to demonstrate the RBP4 levels, association of RBP4 with insulin resistance and influence of testosterone treatment on this cytokine in patients with idiopathic hypogonadotropic hypogonadism.

ELIGIBILITY:
Inclusion Criteria:

decreased serum testosterone concentration below the normal range (serum T < 300ng/dL), FSH and LH levels within or below the normal range, absence of a pituitary or hypothalamic mass lesions on MRI, presence of gonadotropin response to repetitive doses of GnRH, normal smell test and normal karyotypes

Exclusion Criteria:

previous androgen treatment, history of smoking, presence of bilateral anorchia, intellectual deficiency, diabetes mellitus, arterial hypertension or dyslipoproteinemia, medication of any kind and drug abuse. Because of possible confounding effects, patients with other hormone deficiencies were excluded.

-

Ages: 19 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with hypogonadotrophic hypogonadism
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Retinol binding protein 4, hs-CRP levels in patients with idiopathic hypogonadotrophic hypogonadism | 2008-2012

SECONDARY OUTCOMES:
Effect of testosterone treatment on retinol binding globulin 4 and hs-CRP levels in patients with hypogodotrophic hypogonadism | 2008-2012

CONTACTS AND LOCATIONS:
Overall Officials: Aydogan Aydogdu, MD, Study Director — Gulhane School of Medicine, Department of Endocrinology and Metabolism
Locations (1):
- Gulhane School of Medicine Dep. of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)